CLINICAL TRIAL: NCT01408680
Title: Assessing the Effect of the Dietary Supplement Coenzyme Q10 on Biomarkers of Oxidative Stress, Systemic Inflammation, and Endothelial Function in Hemodialysis Patients
Brief Title: CoQ10 Biomarker Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jonathan Himmelfarb, Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 40428-A; R21AT004265 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-08-03 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Oxidative Stress; Inflammation; Endothelial Dysfunction
Keywords: End-stage Renal Disease; Hemodialysis; Cardiovascular Disease; Antioxidants; Atherosclerosis; Coenzyme Q10
MeSH Terms: conditions — Inflammation; Kidney Failure, Chronic; Cardiovascular Diseases; Atherosclerosis | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Coenzyme Q10 600 mg (Active Comparator)
  Interventions: Dietary Supplement: Coenzyme Q10
- Coenzyme Q10 1200 mg (Active Comparator)
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Wafer taken daily by mouth for duration of study, containing Coenzyme Q10 at 600 mg.
  Other Names: CoQ10
  Arms: Coenzyme Q10 600 mg
Dietary Supplement: Coenzyme Q10 — Wafer taken daily by mouth for duration of study, containing Coenzyme Q10 at 1200 mg.
  Other Names: CoQ10
  Arms: Coenzyme Q10 1200 mg
Dietary Supplement: Placebo — Wafer taken daily by mouth for duration of study, containing inactive ingredients. Wafer is indistinguishable from those wafers containing CoQ10.
  Arms: Placebo

SUMMARY:
The investigators believe that relieving the oxidative stress experienced by hemodialysis patients may help improve cardiovascular health.

In this study, the investigators hypothesize that administration of coenzyme Q10, as a targeted antioxidant therapy, will ameliorate the excessive oxidative stress experienced by hemodialysis patients. This will lead to improvements in biomarkers of:

* oxidative stress status
* inflammatory status
* endothelial dysfunction

DETAILED DESCRIPTION:
There are more than 400,000 patients receiving dialysis in the United States, and the investigators expect that this number will go up. For those on hemodialysis, cardiovascular disease (CVD) accounts for a large part of the health problems that these patients have. Cardiovascular problems come from damage to the heart or blood vessels.

At present, the investigators have no treatments proven to help prevent CVD in those on dialysis. For the general population, the investigators know about many factors that increase the risk of CVD, such as having a high level of "bad" cholesterol. But for people on dialysis, the investigators believe that there are other risk factors that are just as important in the development of CVD.

People on dialysis often have high blood levels of waste products. This is called "uremia". The investigators believe that uremia can set up chemical reactions in the blood which can lead to hardening of the arteries (atherosclerosis), an important part of CVD. Compounds called antioxidants, which stop the chemical reactions, may help prevent CVD.

Coenzyme Q10 is a naturally occurring compound in blood and tissues. It is also a readily available dietary supplement often used as an alternative to other medicines. It is a strong antioxidant. The investigators already know that blood levels of coenzyme Q10 are lower in hemodialysis patients. Because of this, it is important for us to find out if giving coenzyme Q10 to hemodialysis patients can help prevent CVD.

In addition, many people take medications called "statins" to help reduce risk for cardiovascular disease. The investigators know that statins can lower coenzyme Q10. It is important for us to know if hemodialysis patients taking statins have lower levels of coenzyme Q10. It may be that taking coenzyme Q10 could increase the good effects of statin medication in hemodialysis patients.

This study will not last long enough for us to look at the development of CVD in subjects. But the investigators will be able to look at biomarkers of oxidative stress, systemic inflammation, and endothelial function. The investigators know that these biomarkers tell us about uremia and other harmful chemical reactions in the blood. If coenzyme Q10 improves the biomarkers, then the investigators believe that it will also help prevent CVD in hemodialysis patients. Our goal is for improvements in cardiovascular risk for those on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease receiving thrice weekly hemodialysis
* Age ≥ 18 or ≤ 85 years
* Life expectancy greater than one year
* Ability to understand and provide informed consent for participation in the study

Exclusion Criteria:

* History of poor adherence to hemodialysis or medical regimen
* Prisoners, patients with significant mental illness, and other vulnerable populations
* AIDS (HIV seropositivity is not an exclusion criteria)
* Active malignancy excluding basal cell carcinoma of the skin
* Gastrointestinal dysfunction requiring parenteral nutrition
* History of functional kidney transplant < 6 months prior to study entry
* Anticipated live donor kidney transplant
* Patients taking vitamin E supplements > 60 IU/day, vitamin C > 150 mg/day or other antioxidant or nutritional supplements
* Incident hemodialysis patients (defined as within 90 days of dialysis initiation)
* Patients hospitalized for more than 5 days within the past 30 days.
* Patients being dialyzed with a tunneled catheter as a temporary vascular access
* Patients with a history of a major atherosclerotic event (defined as combined incidence of myocardial infarction, urgent target-vessel revascularization, coronary bypass surgery, and stroke) within six months
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Oxidative Stress Status at 1 month | 1 month
  We will examine whether administration of coenzyme Q10 will ameliorate the excessive oxidative stress burden as evidenced by changes in serum biomarkers of oxidative stress at the 1-month visit.
Change from Baseline in Oxidative Stress Status at 2 months | 2 months
  We will examine whether administration of coenzyme Q10 will ameliorate the excessive oxidative stress burden as evidenced by changes in serum biomarkers of oxidative stress at the 2-month visit.
Change from Baseline in Oxidative Stress Status at 4 months | 4 months
  We will examine whether administration of coenzyme Q10 will ameliorate the excessive oxidative stress burden as evidenced by changes in serum biomarkers of oxidative stress at the 4-month visit.

SECONDARY OUTCOMES:
Change from Baseline in Inflammatory Status at 1 month | 1 month
  We will examine whether administration of coenzyme Q10 will have an effect on inflammation as evidenced by changes in serum biomarkers of inflammatory status at the 1-month visit.
Change from Baseline in Inflammatory Status at 2 months | 2 months
  We will examine whether administration of coenzyme Q10 will have an effect on inflammation as evidenced by changes in serum biomarkers of inflammatory status at the 2-month visit.
Change from Baseline in Inflammatory Status at 4 months | 4 months
  We will examine whether administration of coenzyme Q10 will have an effect on inflammation as evidenced by changes in serum biomarkers of inflammatory status at the 4-month visit.
Change from Baseline in Endothelial Function at 1 month | 1 month
  We will examine whether administration of coenzyme Q10 will have an effect on endothelial function as evidenced by changes in serum biomarkers and Pulse Amplitude Tonometry scores at the 1-month visit.
Change from Baseline in Endothelial Function at 2 months | 2 months
  We will examine whether administration of coenzyme Q10 will have an effect on endothelial function as evidenced by changes in serum biomarkers and Pulse Amplitude Tonometry scores at the 2-month visit.
Change from Baseline in Endothelial Function at 4 months | 4 months
  We will examine whether administration of coenzyme Q10 will have an effect on endothelial function as evidenced by changes in serum biomarkers and Pulse Amplitude Tonometry scores at the 4-month visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — University of Washington, Kidney Research Institute
Locations (1):
- Northwest Kidney Centers, Seattle, Washington, United States

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- See also: The mission of Northwest Kidney Centers is to promote the optimal health, quality of life and independence of people with kidney disease, through patient care, education and research. — http://www.nwkidney.org/
- See also: The Kidney Research Institute is a collaboration between Northwest Kidney Centers and UW Medicine focused on developing early detection, prevention and treatment of kidney disease and its complications. — http://kri.washington.edu/